CLINICAL TRIAL: NCT00485615
Title: An Open-label, Pilot Study Evaluating the Efficacy of Enteric-coated Eicosapentaenoic Acid (o3mega+Joy) in the Treatment of Social Phobia
Brief Title: An Open Label Trial of Omega 3(o3mega+Joy)in the Treatment of Social Phobia
Acronym: OMEGA3SP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: START Clinic for Mood and Anxiety Disorders (Other)
Collaborators: Genuine Health (Industry)
Responsible Party: Principal Investigator, Dr. Martin A. Katzman, Principal Investigator, START Clinic for Mood and Anxiety Disorders
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHOMEGA3SP
Record Dates: First submitted 2007-06-11; First posted 2007-06-13 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2010-06

CONDITIONS: Social Anxiety Disorder
Keywords: eicosapentaenoic acid; fish oil; Omega 3; Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): OMEGA 3
  Interventions: Drug: Omega 3 Joy enteric coated concentrated fish oil

INTERVENTIONS:
Drug: Omega 3 Joy enteric coated concentrated fish oil — 1500-3000mg; one per day

SUMMARY:
The primary objective is to evaluate the efficacy of an enteric-coated, eicosapentaenoic acid-concentrated fish oil in the treatment of social phobia. A secondary objective is to determine if treatment outcome is related to plasma phospholipid essential fatty acid status, niacin skin flush and measures of lipid/protein peroxidation.

DETAILED DESCRIPTION:
Subjects meeting criteria for Social Anxiety Disorder, will receive enteric-coated, eicosapentaenoic acid-concentrated fish oil (O3mega+Joy) for 12 weeks of treatment for social phobia. A secondary objective is to determine if treatment outcome is related to changes in plasma phospholipid essential fatty acid status, niacin skin flush and measures of lipid/protein change.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for this trial are patients who meet all of the following criteria:

  1. The patient has provided signed informed consent.
  2. Outpatients aged 18-65 (extremes included).
  3. Patients with a primary diagnosis of Social Phobia according to DSM IV (300.23) criteria (diagnosis to be made using the Mini International Neuropsychiatric Interview (MINI)).
  4. On the basis of a physical examination, medical history and basic laboratory screening, the patient is, in the investigators opinion, in a suitable condition.
  5. Willing and able to attend study appointments in the correct time windows.

     Exclusion Criteria:
* Patients meeting one or more of the following criteria cannot be selected for inclusion:

  1. Any other axis I diagnosis that was a primary disorder in the previous six months.
  2. Continuation or commencement of formal psychotherapy.
  3. Alcohol or drug abuse as defined in the DSM IV within the last six months.
  4. Mania or hypomania as defined in the DSM IV.
  5. Current use of or commencement of antidepressant and anxiolytic medications.
  6. Patients who have been on an antidepressant or other anxiolytic prior to the study, will have discontinued it more than two weeks prior to entry into the study. Those who have been on fluoxetine, will have been off of it for at least 5 weeks
  7. Patients who have been on an herbal or alternative treatment judged to be potentially anxiolytic or with psychobiological activity, will have terminated usage of the agent more than two weeks prior to entering the study..
  8. Any psychotic disorder.
  9. Eating disorders as defined in the DSM IV.
  10. Mental retardation or other cognitive disorder.
  11. Clinical interpretation of apparent suicide risk.
  12. Previous treatment efforts using 4000mg or more of fish oil daily.
  13. Current use of or commencement of essential fatty acid supplementation.
  14. Significant alterations from Standard North American Diet ie any special diets either restrictive of or inclusive of typical carbohydrate, protein and fat intake.
  15. Known sensitivity to fish oil or fish products.
  16. Any disorder of clotting or current use of warfarin.
  17. Laboratory values at screening or in medical history that may be considered through clinical interpretation to be significant.
  18. Diseases which could, through clinical interpretation, interfere with the assessments of safety, tolerability and efficacy.
  19. Serious illness: Liver or renal insufficiency, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurological, infectious, neoplastic or metabolic disturbance.
  20. The patient is, in the opinion of the investigator, unlikely to be able to comply with the clinical trial protocol, or is unsuitable for any other reasons.
  21. Pregnant and breastfeeding females
  22. Females of childbearing years who do not use contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Changes in intensity of the vasodilatory response to 10 mM topical m-N over 16 weeks. | Pre treatment - Post treatment

SECONDARY OUTCOMES:
SPIN, SIAS,SPS, ASI, BDI, BAI, SDS, Euroquol, SF 36, BI/BAS, BTSQ, BPS, Niacin Flushing Challenge | Post treatment - Pre Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Katzman, MD, Principal Investigator — START Clinic for Mood and Anxiety Disorders
Locations (1):
- START Clinic for Mood and Anxiety Disorders 900-790 Bay St., Toronto, Ontario, Canada